CLINICAL TRIAL: NCT03579368
Title: A Prospective Evaluation of the Tecnis Symfony Extended Range of Vision Presbyopia Correcting IOL
Brief Title: Prospective Evaluation of the Tecnis Symfony Intraocular Lens (IOL)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kovach Eye Institute (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00025285
Record Dates: First submitted 2018-06-15; First posted 2018-07-06 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-06

CONDITIONS: Cataract; Cataract Senile
Keywords: Cataract; IOL; Presbyopia Correcting IOL; Patient Satisfaction; Spectacle Independence
MeSH Terms: conditions — Cataract; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Single group study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Symfony Implantation (Other): Patients undergoing bilateral IOL implantation with the Tecnis Symfony Extended Range of Vision IOL at a single surgical site
  Interventions: Device: Symfony implantation

INTERVENTIONS:
Device: Symfony implantation — Bilateral Symfony IOL Implantation

SUMMARY:
Advances in cataract surgery and premium IOLs have allowed the ophthalmologist and optometrist to embrace the fact, as with Lasik patients, that refractive cataract surgery can allow their patients to be potentially free or less dependent on glasses. However, fewer than 13% of all patients undergoing cataract surgery today choose a premium IOL and of these approximately 5% are presbyopic IOLs.

The need for greater optometric involvement in cataract surgery is necessary as demand for cataract surgery increases with the population ageing. According to a recent American Optometric Association survey, optometrists diagnose, on average, 13 cases of cataracts per month and refer or co-manage about half of them that are sent for surgery. Since patients base their decision and selection primarily on doctor recommendations, it is incumbent on the optometric community to be well informed on the benefits of the Advanced Technology IOLs.

There is currently no data that has been collected comparing Advanced Technology IOLs and their clinical outcome and acceptance rate among patients co-managed with optometrists. This pilot study will study the subjective visual symptoms, spectacle independence at various distances and patient satisfaction after bilateral implantation of the Tecnis Symfony Extended Range of Vision Advanced Technology IOL in this co-managed care environment. The primary assessment tool will be a Non-directed Patient Satisfaction and Symptoms Questionnaire. Initial questions would include; "How satisfied are you with your spectacle-free vision at distance/intermediate/near?", "Would you choose the same lens again?" and "Would you recommend the same lens to your relatives and friends". Similarly, with regard to Photic phenomena / visual symptoms, we would ask "Do you experience any problems with your vision?" and only follow up with specific questions on severity once the patient volunteers a specific symptom..

The surgery form will include a question determining the surgeon's satisfaction with the individual Symfony lens implantation. At last visit the optometric investigator will be asked about his satisfaction with the performance of the Symfony lens. This will allow monitoring of any progression of satisfaction as more experience with the lens is obtained.

DETAILED DESCRIPTION:
Symfony Extended Range of Vision IOL was approved by the FDA for commercial use in the United States in August 2016 demonstrating reasonable assurance of safety and effectiveness (PMA # P980040 S065). The Symfony IOL diffracts light in a way that allows an extended range of focus, rather than focusing light at distinct points. Monofocal IOLs have one distinct focus, which can be set by the surgeon for distance, intermediate, or near. Multifocal IOLs have two distinct foci for light, at distance and intermediate or near. The proposed optics of the Symfony are geared toward elongating the eye's focus, rather than producing two distinct focal points. This elongated focus allows a more continuous spectrum of sharp vision from distance through intermediate and to near points. Additionally, because light is not focused at two distinct points, glare and halos should not be as noticeable.

The Symfony IOL offers many advantages to patients, including the absence of a blurry zone of vision between two distinct focal points. With this comes the possibility of reduced glare and halos. Additionally, the extended depth of focus, which is more consistent with accommodating lenses, is not dependent on postoperative movement of the IOL.

An important consideration when selecting this lens is the patient's desired quality of near vision. The defocus curve of the Symfony lens shows vision between 20/15 and 20/20 from distance to approximately 66 cm (2 ft). Vision ranges from 20/20 to 20/30 in the intermediate range of vision until about 50 cm (19 in) and then drops to 20/40 at 40 cm (1 ft). For patients looking for crisp vision for close reading, this lens may not meet expectations.

This study will simply involve following patients who are implanted with the Tecnis Symfony Extended Range of Vision IOL. No clinical testing will be performed on the patients other than those routinely performed by the examining clinician. The only non-routine aspect to the study is the administration of questionnaires to evaluate symptoms and satisfaction. Thus it appears that this study introduces no extra risk to the patient over and above that of the underlying cataract surgery.

The objectives of this single surgical site clinical study are to study the subjective visual symptoms, spectacle independence at various distances and patient satisfaction after bilateral implantation of the Tecnis Symfony Extended Range of Vision IOL in a co-managed care environment (Ophthalmologists and Optometrists).

The patient population for this clinical study will be 200 bilaterally implanted Symfony IOL patients from 10 optometric practices who fit the inclusion/exclusion criteria for this study determined at 1 month postoperatively and were referred to a single surgical site.

This study will be a prospective clinical investigation. The study endpoint will be at 3 months postoperatively. Subjects will be recruited from the referring optometrist's current patient population. Subjects will be enrolled into the study in a sequential manner only after it has been determined that they are qualified according to the Clinical Protocol inclusion and exclusion criteria. The study will involve a single surgical site (Principal Investigator and Surgeon Co-Investigator) and 10 co-managing optometric referring sites (Co-Investigators). Informed consent, testing study subject questionnaire administration will be conducted at the co-managing optometric sites. Surgery will be performed at the single surgical site.

The incidence of subjective visual symptoms, spectacle independence at various distances and patient satisfaction will be tabulated for each center and for the population as a whole

ELIGIBILITY:
Inclusion Criteria:

* Patients bilaterally implanted with the Tecnis® Symfony Extended Range of Vision IOL
* Age 18 and older
* Patient targeted for emmetropic refraction both eyes (OU)
* Postoperative refractive spherical equivalent within ± 0.5 Diopters OU
* Postoperative refractive cylinder of ≤ 0.75 Diopters OU
* Clear intraocular media
* Availability, willingness and sufficient cognitive awareness to comply with examination procedures
* Subjects must have best corrected visual acuity (BCDVA) better than 20/30 after cataract removal and IOL implantation OU

Exclusion Criteria:

* Acute or chronic diseases or illness that would increase risk or confound study results, such as proliferative or moderate to severe background diabetic retinopathy, macular degeneration, or cystoid macular edema.
* Subjects with any anterior pathology that would be likely to increase the risk of complications from cataract and IOL surgery such as keratoconus, Fuchs dystrophy or any other previous serious corneal disease, pupil irregularity, unmanaged (severe) dry eyes, ocular infection or inflammation or uncontrolled glaucoma.
* Subjects with associated ocular conditions that could affect the stability of the IOL such as zonular dialysis or pseudoexfoliation syndrome.
* Subjects with central nervous system or motility issue such as dementia or alternating mono-fixators, e.g. amblyopia or strabismus
* Subjects with intra-operative complications such as posterior capsule rupture, or other unresolved complications affecting visual outcome
* History of any refractive or intraocular surgery (not including treatment for retinal holes)
* Clinically significant Ptosis
* Pupil abnormalities (non-reactive, tonic, abnormally shaped pupils, or pupils that do not dilate at least 3.5mm under mesopic/scotopic conditions)
* Patient participation in another clinical trial (former participation is no exclusion criterion)
* Use of systemic or ocular medication that might affect vision
* Patients whose primary visual requirement postoperatively is crisp, clear uncorrected visual acuity for near distances at less than 20 inches.
* Active ocular surface disease affecting the refractive surface properties of the cornea (i.e. Meibomian gland dysfunction, or moderate to severe dry eye etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-07-05 (Estimated); Primary Completion 2019-04-15 (Estimated); Study Completion 2019-05-15 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction & Spectacle independence | 3 months postoperatively
  Patient questionaire

SECONDARY OUTCOMES:
Patient satisfaction & Spectacle independence | 1 month postoperatively
  Patient questionaire
Surgeon Satisfaction | Intraoperative
  Satisfaction questionaire
Referring Optometrist Satisfaction | 3 months postoperatively
  Satisfaction questionaire
Patient Symptoms | 1 month postoperative
  Symptom Questionaire
Patient Symptoms | 3 months postoperative
  Symptom Questionaire
Adverse Events and Complications | 1 month postoperative
  Adverse Events and Complications
Adverse Events and Complications | 3 months postoperative
  Adverse Events and Complications

CONTACTS AND LOCATIONS:
Overall Officials: Donald R Sanders, Study Director — Center for Clinical Research

IPD SHARING:
Plan to Share IPD: No